CLINICAL TRIAL: NCT01063179
Title: A PHASE III, MULTI-CENTER, RANDOMIZED OPEN LABEL STUDY OF VELCADE, MELPHALAN, PREDNISONE AND THALIDOMIDE (V-MPT) Versus VELCADE, MELPHALAN, PREDNISONE (V-MP) IN ELDERLY UNTREATED MULTIPLE MYELOMA PATIENTS
Brief Title: Velcade, Melphalan, Prednisone And Thalidomide Versus Velcade, Melphalan, Prednisone in Multiple Myeloma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIMEMA-MM-03-05; 2005-004745-33 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma
Keywords: Elderly patients; Bortezomib; Thalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone; Thalidomide; VMP regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: VMPT (Experimental): Induction therapy with nine 5-week courses of VELCADE/Melphalan/Prednisone/Thalidomide (V-MPT) followed by maintenance therapy with Thalidomide and VELCADE
  Interventions: Drug: Bortezomib, Melphalan, Prednisone, Thalidomide
- VMP (Active Comparator): Induction therapy with nine 5-week courses of either VELCADE/Melphalan/Prednisone (V-MP).
  No maintenance is scheduled.
  Interventions: Drug: Bortezomib, Melphalan, Prednisone

INTERVENTIONS:
Drug: Bortezomib, Melphalan, Prednisone, Thalidomide — Induction therapy:
  9 courses with weekly VELCADE (4 doses) in combination with oral Melphalan 9 mg/m2,oral Prednisone 60 mg/m2 once daily on Days 1 to 4 of each course and Thalidomide 50 mg/day continuously. The dose of VELCADE is 1.3 mg/m2 administered as a bolus IV injection, on days 1, 8, 15, 22.
  Maintenance therapy:
  Thalidomide 50 mg/day continuously in combination with VELCADE 1.3 mg or maximum dose tolerated/m2/2 weeks. The maintenance will be initiated at the end of the 9th course and will be stopped after progression. The median expected duration of the maintenance treatment is approximately 2 years.
  Other Names: Bortezomib; Velcade; Thalidomide
  Arms: Arm A: VMPT
Drug: Bortezomib, Melphalan, Prednisone — Induction therapy: 9 courses with weekly VELCADE(4 doses) in combination with oral Melphalan 9 mg/m2 and oral Prednisone 60 mg/m2 once daily on Days 1 to 4 of each course. No maintenance therapy is scheduled
  Other Names: Boirtezomib; velcade
  Arms: VMP

SUMMARY:
The proposed study will evaluate whether the combination of VELCADE, Thalidomide , Melphalan and Prednisone (V-MPT), as induction treatment for newly diagnosed elderly MM patients, improves outcomes compared to the combination VELCADE-MP.

DETAILED DESCRIPTION:
This phase III study represents a prospective randomized open label multicenter trial to evaluate whether the combination of VELCADE, Melphalan, Prednisone and Thalidomide (V-MPT), as induction treatment for newly diagnosed elderly MM patients, improves outcomes compared to the combination VELCADE-MP.

Subjects will be randomized in a 1:1 allocation between:

Arm A: 250 patients: V-MPT treatment Arm B: 250 patients: V-MP treatment Patients excluded from randomization are to be registered in Arm C. Patients randomized in arm A (Thalidomide based) will be further enrolled in the sub-study about the DVT prophylaxis.

Patients will be evaluated at scheduled visits in up to 3 study periods: pre-treatment, treatment and long-term follow-up (LTFU).

1. Pre-treatment period:

   Screening visits, performed at study entry. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility After registration subjects will be randomized.
2. Treatment period:

   Subjects in Arm A will receive:
   1. Induction therapy:

      nine 5-week courses of VELCADE/Melphalan/Prednisone/Thalidomide (V-MPT)
   2. Maintenance therapy:

   Thalidomide in combination with VELCADE

   Subjects in Arm B will receive:
   1. Induction therapy:

      nine 5-week courses of VELCADE/Melphalan/Prednisone (V-MP)
   2. No maintenance therapy is scheduled At the end of induction treatment or at the time of discontinuation of all study drugs, all patients are to attend study center visits on an every 6 to 8-week basis, until development of confirmed Progressive Disease (PD)
3. LTFU period:

After development of confirmed PD all patients are to be followed for survival every 3 months via telephone or office visit.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 year old and not a candidate for stem cell transplant, or younger who refuses or is not eligible for high-dose therapy
* Symptomatic multiple myeloma or asymptomatic multiple myeloma with related organ or tissue damage
* Presence of measurable disease
* Karnofsky performance status (PS) > 60%
* Able to read and complete the HRQOL instruments
* Agrees to use an acceptable barrier method for contraception for the duration of the study
* Pretreatment clinical laboratory values within 14 days of randomization:

platelet count ≥ 100x109/L

* hemoglobin ≥ 8 g/dL
* absolute neutrophil count (ANC) ≥ 1.0x109/L
* AST ≤ 2.5 times the upper limit of normal
* ALT ≤ 2.5 times the upper limit of normal
* total bilirubin ≤ 1.5 times the upper limit of normal
* serum creatinine ≤ 2.5mg/dL
* corrected serum calcium <14 mg/dL (<3.5 mmol/L)
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Women of child-bearing potential must agree to use 2 methods of contraception: 1 effective (for example hormonal or tubal ligation) and 1 barrier (for example latex condom, diaphragm) for at least 4 weeks before starting the therapy, during the Treatment Period, and for 4 weeks after the last dose;
* Males must agree to use barrier contraception (latex condoms) when engaging in reproductive activity during the Treatment Period and for 4 weeks after the last dose.

Exclusion Criteria:

* Diagnosis of smoldering multiple myeloma or MGUS.
* Diagnosis of Waldenstrom's disease
* Prior or current systemic therapy for multiple myeloma including steroids (with exception of emergency use of a short course [maximum 4 days] of steroids before randomization or prior or current use of biphosphonates)
* Radiation therapy within 30 days before randomization
* Plasmapheresis within 30 days before randomization
* Major surgery within 30 days before randomization (Kyphoplasty is not considered major surgery)
* History of allergic reaction attributable to compounds containing boron or mannitol, or to Thalidomide
* Peripheral neuropathy Grade 2 or higher, as defined by National Cancer Institute Common Toxicity Criteria (NCI CTC) 3.0
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
* Other malignancy within the past 5 years. Exceptions: basal cell or non metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or FIGO Stage 1 carcinoma of the cervix
* Concurrent medical condition or disease (e.g., active systemic infection, uncontrolled diabetes, pulmonary disease) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study
* Use of any investigational drugs within 30 days before randomization.
* Pregnant or lactating women. A serum β-hCG pregnancy test must be performed at the Screening visit, for female patients of child-bearing potential. If the test is positive, the patient must be excluded from the study. Confirmation that the patient is not pregnant must be established by a negative serum or urinary pregnancy test with the result obtained 1 day prior to the Baseline visit (or the day of the visit if results are available before drug delivery).

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 511 (Actual)
Dates: Start 2006-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Determine whether the V-MPT combination improves progression free survival (PFS) | Approximately 24 months

SECONDARY OUTCOMES:
Determine whether the VMPT combination improves:Response rate, Overall Survival rate, Time and duration of response, Assess the safety, Assess the prognostic factors | Approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mario Boccadoro, MD, Principal Investigator — Divisione di Ematologia dell'Università di Torino, A.O.U. S. Giovanni Battista, Torino;Italy
Locations (1):
- A.O.U. S. Giovanni Battista, Torino, Italy

REFERENCES:
- [Derived] Larocca A, Mina R, Offidani M, Liberati AM, Ledda A, Patriarca F, Evangelista A, Spada S, Benevolo G, Oddolo D, Innao V, Cangiolosi C, Bernardini A, Musto P, Amico V, Fraticelli V, Paris L, Giuliani N, Falcone AP, Zambello R, De Paoli L, Romano A, Palumbo A, Montefusco V, Hajek R, Boccadoro M, Bringhen S. First-line therapy with either bortezomib-melphalan-prednisone or lenalidomide-dexamethasone followed by lenalidomide for transplant-ineligible multiple myeloma patients: a pooled analysis of two randomized trials. Haematologica. 2020 Apr;105(4):1074-1080. doi: 10.3324/haematol.2019.220657. Epub 2019 Jun 27. PMID 31248973
- [Derived] Montefusco V, Gay F, Spada S, De Paoli L, Di Raimondo F, Ribolla R, Musolino C, Patriarca F, Musto P, Galieni P, Ballanti S, Nozzoli C, Cascavilla N, Ben-Yehuda D, Nagler A, Hajek R, Offidani M, Liberati AM, Sonneveld P, Cavo M, Corradini P, Boccadoro M. Outcome of paraosseous extra-medullary disease in newly diagnosed multiple myeloma patients treated with new drugs. Haematologica. 2020 Jan;105(1):193-200. doi: 10.3324/haematol.2019.219139. Epub 2019 Jun 20. PMID 31221778
- [Derived] Saltarella I, Morabito F, Giuliani N, Terragna C, Omede P, Palumbo A, Bringhen S, De Paoli L, Martino E, Larocca A, Offidani M, Patriarca F, Nozzoli C, Guglielmelli T, Benevolo G, Callea V, Baldini L, Grasso M, Leonardi G, Rizzo M, Falcone AP, Gottardi D, Montefusco V, Musto P, Petrucci MT, Dammacco F, Boccadoro M, Vacca A, Ria R. Prognostic or predictive value of circulating cytokines and angiogenic factors for initial treatment of multiple myeloma in the GIMEMA MM0305 randomized controlled trial. J Hematol Oncol. 2019 Jan 9;12(1):4. doi: 10.1186/s13045-018-0691-4. PMID 30626425
- [Derived] Cerrato C, Di Raimondo F, De Paoli L, Spada S, Patriarca F, Crippa C, Mina R, Guglielmelli T, Ben-Yehuda D, Oddolo D, Nozzoli C, Angelucci E, Cascavilla N, Rizzi R, Rocco S, Baldini L, Ponticelli E, Marcatti M, Cangialosi C, Caravita T, Benevolo G, Ria R, Nagler A, Musto P, Tacchetti P, Corradini P, Offidani M, Palumbo A, Petrucci MT, Boccadoro M, Gay F. Maintenance in myeloma patients achieving complete response after upfront therapy: a pooled analysis. J Cancer Res Clin Oncol. 2018 Jul;144(7):1357-1366. doi: 10.1007/s00432-018-2641-5. Epub 2018 Apr 19. PMID 29675792
- [Derived] Caltagirone S, Ruggeri M, Aschero S, Gilestro M, Oddolo D, Gay F, Bringhen S, Musolino C, Baldini L, Musto P, Petrucci MT, Gaidano G, Passera R, Bruno B, Palumbo A, Boccadoro M, Omede P. Chromosome 1 abnormalities in elderly patients with newly diagnosed multiple myeloma treated with novel therapies. Haematologica. 2014 Oct;99(10):1611-7. doi: 10.3324/haematol.2014.103853. Epub 2014 Jul 11. PMID 25015938
- [Derived] Palumbo A, Bringhen S, Larocca A, Rossi D, Di Raimondo F, Magarotto V, Patriarca F, Levi A, Benevolo G, Vincelli ID, Grasso M, Franceschini L, Gottardi D, Zambello R, Montefusco V, Falcone AP, Omede P, Marasca R, Morabito F, Mina R, Guglielmelli T, Nozzoli C, Passera R, Gaidano G, Offidani M, Ria R, Petrucci MT, Musto P, Boccadoro M, Cavo M. Bortezomib-melphalan-prednisone-thalidomide followed by maintenance with bortezomib-thalidomide compared with bortezomib-melphalan-prednisone for initial treatment of multiple myeloma: updated follow-up and improved survival. J Clin Oncol. 2014 Mar 1;32(7):634-40. doi: 10.1200/JCO.2013.52.0023. Epub 2014 Jan 21. PMID 24449241
- [Derived] Morabito F, Gentile M, Mazzone C, Rossi D, Di Raimondo F, Bringhen S, Ria R, Offidani M, Patriarca F, Nozzoli C, Petrucci MT, Benevolo G, Vincelli I, Guglielmelli T, Grasso M, Marasca R, Baldini L, Montefusco V, Musto P, Cascavilla N, Majolino I, Musolino C, Cavo M, Boccadoro M, Palumbo A. Safety and efficacy of bortezomib-melphalan-prednisone-thalidomide followed by bortezomib-thalidomide maintenance (VMPT-VT) versus bortezomib-melphalan-prednisone (VMP) in untreated multiple myeloma patients with renal impairment. Blood. 2011 Nov 24;118(22):5759-66. doi: 10.1182/blood-2011-05-353995. Epub 2011 Sep 27. PMID 21951682
- [Derived] Gay F, Larocca A, Wijermans P, Cavallo F, Rossi D, Schaafsma R, Genuardi M, Romano A, Liberati AM, Siniscalchi A, Petrucci MT, Nozzoli C, Patriarca F, Offidani M, Ria R, Omede P, Bruno B, Passera R, Musto P, Boccadoro M, Sonneveld P, Palumbo A. Complete response correlates with long-term progression-free and overall survival in elderly myeloma treated with novel agents: analysis of 1175 patients. Blood. 2011 Mar 17;117(11):3025-31. doi: 10.1182/blood-2010-09-307645. Epub 2011 Jan 12. PMID 21228328
- [Derived] Bringhen S, Larocca A, Rossi D, Cavalli M, Genuardi M, Ria R, Gentili S, Patriarca F, Nozzoli C, Levi A, Guglielmelli T, Benevolo G, Callea V, Rizzo V, Cangialosi C, Musto P, De Rosa L, Liberati AM, Grasso M, Falcone AP, Evangelista A, Cavo M, Gaidano G, Boccadoro M, Palumbo A. Efficacy and safety of once-weekly bortezomib in multiple myeloma patients. Blood. 2010 Dec 2;116(23):4745-53. doi: 10.1182/blood-2010-07-294983. Epub 2010 Aug 31. PMID 20807892